CLINICAL TRIAL: NCT07344896
Title: Effects of a Mindfulness-Based Stress Reduction Program on Aging Anxiety and Body Image in Middle-Aged Women: A Randomized Controlled Trial
Brief Title: MBSR Effects on Aging Anxiety and Body Image
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: KTO Karatay University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Karatay University
Record Dates: First submitted 2025-12-08; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2025-12

CONDITIONS: Body Image; Mindfulness Based Stress Reduction; Middle Aged
Keywords: aging anxiety; middle age woman; mindfulness; body image

STUDY DESIGN:
Intervention Model Description: In this study, block randomization will be applied. Participants will be stratified based on two variables: menopausal status (yes/no) with two levels, and educational level (literate-primary school / high school / university and above) with three levels. Within each stratum, block randomization will be conducted using variable block sizes (4 and 6) to ensure a 1:1 allocation ratio.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mindfulness-based stress reduction program intervention group (Experimental): After the pre-test, a mindfulness-based stress reduction program will be implemented. It will be evaluated with a post-test.
  Interventions: Behavioral: bilinçli farkındalık temelli stres azaltma programı
- control group (No Intervention): A pre-test will be administered. No practice will be conducted. Students will be evaluated with a post-test

INTERVENTIONS:
Behavioral: bilinçli farkındalık temelli stres azaltma programı — Following application to the center, the Mindfulness-Based Stress Reduction (MBSR) program will be implemented starting from the scheduled date. The program will last a total of 8 weeks, with one session per week, each session lasting approximately 2 hours. At the end of the 6th week, one day will be designated as a "day of silence," during which a 6-hour session will be conducted.
  The 8-week program is structured around the themes of aging anxiety and body image. During the day of silent awareness (after the 6th week), the 6-hour silence period will include body scan practices, mindful walking, and breathing meditation. The aim of this silent retreat day is to deepen participants' internal awareness.
  Arms: mindfulness-based stress reduction program intervention group

SUMMARY:
This study was designed to determine the effect of a mindfulness-based stress reduction (MBSR) program on aging anxiety and body image among middle-aged women. The primary hypotheses to be tested are as follows:

H0a: There is no difference in the mean scores of the Aging Anxiety Scale between the women in the experimental group who receive the mindfulness-based stress reduction program and the women in the control group.

H0b: There is no difference in the mean scores of the Body Image Scale between the women in the experimental group who receive the mindfulness-based stress reduction program and the women in the control group.

H0c: There is no difference between the pre-intervention and post-intervention mean scores of the Aging Anxiety Scale among the women in the experimental group who receive the mindfulness-based stress reduction program.

H0d: There is no difference between the pre-intervention and post-intervention mean scores of the Body Image Scale among the women in the experimental group who receive the mindfulness-based stress reduction program.

The researchers will compare the experimental group with the control group in order to assess the effect of the mindfulness-based stress reduction program on aging anxiety and body image among middle-aged women.

Participants:

* They will attend an 8-session mindfulness-based stress reduction program.
* They will participate in one silent mindfulness retreat session.

ELIGIBILITY:
Inclusion Criteria:

* At least primary school graduate,
* Being between 45-59 years old,
* Living in Çumra district center,
* Being open to communication and cooperation

Exclusion Criteria:

* Those with chronic illnesses (self-report)
* Foreign nationals Those with psychiatric illnesses (self-report) Those with physical disabilities and limited mobility

Ages: 45 Years to 59 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 58 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Change in Aging Anxiety Score as Measured by the Aging Anxiety Scale for Middle-Aged Women | Baseline and immediately post-intervention (8 weeks)
  Aging anxiety will be assessed using the Aging Anxiety Scale for Middle-Aged Women, a self-report questionnaire consisting of Likert-type items. The outcome will be evaluated as the mean change in total scale score from baseline to immediately post-intervention. Higher scores indicate higher levels of aging anxiety.

SECONDARY OUTCOMES:
Change in Body Image Score as Measured by the Body Image Scale | Baseline and post-intervention (8 weeks)
  Body image will be assessed using the Body Image Scale, a self-report instrument measuring individuals' perceptions and attitudes toward their own bodies. The outcome will be evaluated as the mean change in total scale score from baseline to post-intervention. Higher scores indicate a more positive body image.

CONTACTS AND LOCATIONS:
Overall Officials: Necibe Ş TUNALI, 1, Study Director — KTO KARATAY UNİVERSİTY

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to the sensitive nature of the psychological and health-related information collected from middle-aged women. The dataset includes identifiable variables related to aging anxiety, body image, and mindfulness-based intervention outcomes. Sharing such data may pose confidentiality risks despite anonymization efforts. Aggregated results will be available upon request.

REFERENCES:
- [Background] Aydın, A., & Kabasakal, E. (2022). Turkish adaptation of the Aging Anxiety Scale for middle-aged women: Validity and reliability study. Journal of Basic and Clinical Health Sciences, 6, 173-180. https://doi.org/10.30621/jbachs.2022.1012 Bergman, Y. S., & Segel-Karpas, D. (2018). Future time perspective, loneliness, and depressive symptoms among middle-aged adults: A mediation model. Journal of Affective Disorders, 241, 173-175. https://doi.org/10.1016/j.jad.2018.08.019 Bergman, Y. S., & Segel-Karpas, D. (2021). Aging anxiety, loneliness, and depressive symptoms among middle-aged adults: The moderating role of ageism. Journal of Affective Disorders, 290, 89-92. https://doi.org/10.1016/j.jad.2021.04.077 Cameron, E., Ward, P., Mandville-Anstey, S. A., & Coombs, A. (2018). The female aging body: A systematic review of female perspectives on aging, health, and body image. Journal of Women & Aging, 31(1), 3-17. https://doi.org/10.1080/08952841.2018.1449586 Creswell, J. D. (2017). Mindfulness interventions. Annual Review of Psychology, 68, 491-516. https://doi.org/10.1146/annurev-psych-042716-051139 Fernandez-Jimenez, C., Alvarez-Hernandez, J. F., Salguero-Garcia, D., Aguilar-Parra, J. M., & Trigueros, R. (2020). Validation of the Lasher and Faulkender Anxiety about Aging Scale (AAS) for the Spanish context. International Journal of Environmental Research and Public Health, 17(12), 4231. https://doi.org/10.3390/ijerph17124231 Gendron, T. L., Inker, J. K., Andricosky, R., & Zanjani, F. (2020). Development of the relational ageism scale: Confirmatory test on survey data. International Journal of Aging and Human Development, 90(3), 281-296. https://doi.org/10.1177/0091415019836956 Lee, H., & You, M. (2019). Development of an aging anxiety scale for middle-aged women. Journal of Korean Academy of Nursing, 49(1), 14-25. https://doi.org/10.4040/jkan.2019.49.1.14